CLINICAL TRIAL: NCT07171645
Title: Gender-Affirming Care and Mental Health (GLOW): A Longitudinal Study On Quality of Life, Work Life, and Healthcare Outcomes
Brief Title: Gender-Affirming Care and Mental Health
Acronym: GLOW
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-07577-01
Record Dates: First submitted 2025-08-10; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Gender Dysphoria, Adult; Psychiatric Comorbidities
Keywords: gender dysphoria; self-concept; National Highly Specialized Care (NHV); Identity; Stigma; Mixed Methods
MeSH Terms: conditions — Gender Dysphoria; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with gender dysphoria: The study cohort consists of adults (18+) with gender dysphoria who have been referred to the National Highly Specialized Care Unit (Nationell Högspecialiserad Vård, NHV) for gender dysphoria at Region Skåne, Sweden. This unit serves as one of the national centers for the assessment and treatment of individuals seeking gender-affirming care. Participants are recruited at the initiation of their clinical assessment-a standardized, multidisciplinary evaluation process typically involving psychiatrists, psychologists, and counselors, which spans approximately three months. This assessment constitutes the first formal step toward potential access to gender-affirming interventions.
  Interventions: Other: Assessment regarding gender-affirming care
- Randomized comparison group: A matched randomized comparison group drawn from registries. This group will be used as a comparison for the registry data only.

INTERVENTIONS:
Other: Assessment regarding gender-affirming care — No comparison
  Groups: Individuals with gender dysphoria

SUMMARY:
Introduction Gender-Affirming Care and Mental Health (GLOW) investigates the psychological, medical, and social factors that influence the outcomes of gender-affirming care, as well as its impact on mental health, work capacity, and quality of life. Gender dysphoria is defined as the incongruence of a person's experienced gender and sex assigned at birth. In Sweden, the prevalence of gender dysphoria has increased significantly in recent decades. Still there is no consensus on the long-term outcomes of gender-affirming care.

1. What are the baseline characteristics in individuals seeking gender-affirming care and do any of these predict outcomes of gender-affirmative care?
2. Do individuals with gender dysphoria experience improved or reduced quality of life, gender congruence, or functional capacity after gender-affirming care?
3. Does gender-affirming care reduce or increase psychiatric symptoms and self-concept clarity?
4. What are the effects of gender-affirming care on mortality, work capacity, and healthcare resource utilization as compared to an age and gender matched control group?

Data and Method GLOW targets patients at the Gender Dysphoria Clinic, Region Skåne a National Highly Specialized Care unit (NHV). Mixed methods will be used to analyze data from national registries and self-reported assessments.The NHV status ensures standardized high-quality data collection and clinical follow-up, making this project a unique opportunity to evaluate the care given to individuals with gender dysphoria.

Societal Relevance and Utility The growing demand for gender-affirming care underscores the need for research to identify the most effective interventions. The results may also help reduce stigma and improve social integration for individuals with gender dysphoria.

DETAILED DESCRIPTION:
The GLOW study is a longitudinal investigation designed to evaluate the effects of gender-affirming care on the well-being of individuals diagnosed with gender dysphoria in Sweden. Grounded in an interdisciplinary framework, the study adopts a mixed-methods approach to integrate quantitative registry data and longitudinal self-assessments with in-depth qualitative interviews. This design allows for anunderstanding of the medical, psychological, and social dimensions of gender-affirming care beyond the limitations of cross-sectional studies.

The project is embedded in Region Skåne's National Highly Specialized Care (NHV) unit, ensuring standardized data collection and uniform clinical procedures across participants. Thus, the study benefits from a stable clinical infrastructure and reliable access to a diverse cohort undergoing gender-affirming assessment and treatment. In addition, national health and population registries provide extensive data for long-term follow-up, including health service utilization, prescription records, socio-economic indicators, and mortality data.

GLOW is commited to a collaborative research practice. The project actively involves key stakeholders-healthcare professionals, policymakers, and patient advocacy groups such as Transammans and RFSL. Their input ensures that the study remains aligned with real-world clinical needs and community priorities, enhancing its relevance.

The study is conceptually anchored in the Biopsychosocial Model and draws on Minority Stress Theory, Self-Concept Clarity Theory, and Gender Affirmation Theory. These frameworks support the exploration of how social stressors, identity development, and access to affirming care interact to shape mental health trajectories. This theoretical integration provides a solid foundation for interpreting variability in treatment response and quality-of-life outcomes.

Statistical modeling will be employed to complement traditional analyses, offering probabilistic interpretations and greater flexibility in handling complex longitudinal data structures. Qualitative interviews will be analyzed using thematic methods, with findings triangulated against quantitative trends to increase the validity and depth of insights.

While many existing studies on gender-affirming care focus on short-term or medical outcomes, GLOW takes a broader and longer-term perspective. It includes economic implications, healthcare resource use, work life outcomes, and subjective experiences of identity and social integration. This holistic approach will generate knowledge applicable to clinical care, policy formulation, and public health planning.

Finally, the project emphasizes sustainability. Infrastructure and data collection protocols have been designed to support extended follow-up. In doing so, GLOW aims to contribute not only to scientific literature but also to the development of evidence-based guidelines and inclusive healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 18 years and older.

Referred to the National Highly Specialized Care Unit (NHV) for gender dysphoria at Region Skåne.

Presenting for initial clinical assessment for gender-affirming care.

Able to provide informed consent for participation in the self-report portion of the study.

Participants may identify as female, male, or another gender identity.

Exclusion Criteria:

Inability to read or write Swedish, as all self-report measures and consent forms are in Swedish.

Individuals with protected (secret) identities, such as those under special confidentiality protections or in high-security identity protection programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults (18 years and older) diagnosed with gender dysphoria who have been referred to the National Highly Specialized Care (NHV) Unit for gender dysphoria at Region Skåne. This clinic is one of Sweden's national centers for gender-affirming care, receiving approximately 350-400 new referrals annually. Participants are enrolled at the start of their initial clinical assessment, which is the gateway to potential interventions such as hormone therapy, surgery, voice therapy, and psychological support. The study includes individuals of all gender identities (e.g., female, male, nonbinary) to reflect the diversity of the transgender population. Participants are followed longitudinally using self-report questionnaires, clinical records, and national registry data to assess mental health, identity development, and quality-of-life outcomes across time.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2032-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) to evaluate general health status and functioning.
  Score is converted to a 0-100 scale, where a higher score indicates greater disability or limitation in functioning.

OTHER OUTCOMES:
Generic quality of life | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Measured with EuroQoL-5 Dimension Questionnaire (EQ-5D)
  Describes five levels of problems ("no, mild, moderate, severe, extreme problem") and a scale that typically ranges from 0 ("worst imaginable health") to 100 ("best imaginable health").
Substance Use | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Instruments: Alcohol Use Disorders Identification Test (AUDIT).
  AUDIT produces a score from 0 to 40, with higher scores indicating a greater likelihood of hazardous, harmful, or dependent drinking.
Substance Use | Time Frame: Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Measured using the Drug Use Disorders Identification Test (DUDIT). DUDIT produces a score from 0 to 44, with higher scores indicating more severe drug-related problems or potential dependence.
Self-Concept Clarity and Identity Functioning | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Measured via the Self-Concept and Identity Measure (SCIM) and Level of Personality Functioning Scale - Brief Form 2.0 (LPFS 2).
  SCIM has a total score range from 36 to 180, with higher scores indicating greater identity disturbance,
  LPFS has a range of 12 to 48, where a higher score indicates greater dysfunction.
Change in Mental Health Symptoms | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Measured using the Generalized Anxiety Disorder Scale (GAD-7). The range of GAD 7 is 0 to 21. Higher scores indicate greater severity of anxiety symptoms.
Change in Mental Health Symptoms | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Questions regarding number of suicidal behavior.
Gender Congruence and Life Satisfaction | Baseline, after assessment completion (an average of 1 year), 24 months, and 60 months.
  Measured using the Gender Congruence Life Satisfaction Scale (GCLS).
  Range is 0 to 50. A higher score indicates a more positive outcome (higher gender congruence, better gender-related mental well-being, and better general life satisfaction).
Mortality | 60 months
  Source: Cause of Death Register (CDR)
Work Capacity and Socioeconomic Participation | Baseline and 60 months
  Derived from the Longitudinal Integration Database for Health Insurance and Labour Market Studies (LISA), including employment status and income.
Healthcare Utilization | Baseline and 60 months.
  Source: National Patient Register (NPR)
  Metrics: Number of hospital visits.
Healthcare Utilization | Baseline and 60 months.
  Source: Prescribed Drug Register
  Metrics: Use of medications (number of doses)
Healthcare Utilization | Baseline and 60 months.
  Source: National Patient Register (NPR)
  Metrics: Psychiatric diagnoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Department/Office of Psychiatry, National specialized medical care, Skåne University Hospital, Lund, Sweden., Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided